CLINICAL TRIAL: NCT02055924
Title: A Phase Ib Study of Ibrutinib Combined With R-DHAP or R-DHAOx in Patients With B-cell Lymphomas
Brief Title: Bruton's Tyrosine Kinase (BTK) Inhibition in B-cell Lymphomas
Acronym: BIBLOS
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: ANSM decision due to veino occlusive disease (security alert)
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIBLOS
Record Dates: First submitted 2014-01-31; First posted 2014-02-05 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: B-cell Lymphoma
Keywords: Bruton's tyrosine kinase (BTK) Inhibition in B-cell Lymphomas
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib and immunochemotherapies (Experimental): Combination of immunochemotherapies (R-DHAP or R-DHAOx) and ibrutinib
  Interventions: Drug: Ibrutinib and immunochemotherapies

INTERVENTIONS:
Drug: Ibrutinib and immunochemotherapies — Combination of immunochemotherapies (R-DHAP or R-DHAOx) and ibrutinib
  Other Names: Ibrutinib + R-DHAP; Ibrutinib + R-DHAOx

SUMMARY:
This is an open label, multicenter, dose escalation, phase Ib study to determine the recommended dose by assessing the maximum tolerated dose (MTD), safety and efficacy of ibrutinib in combination with R-DHAP (Group A/Abis) or R-DHAOx (Group B/Bbis) for patients with B-cell malignancies. This dose escalation will be followed by an exploratory expansion phase in 3 groups of 12 patients each (Group A/Abis, Group B/B bis and Group C).

During Part 1 Dose Escalation, the "3+3" design will be applied. Three doses of ibrutinib (280, 420 and 560 mg) will be examined sequentially in each cohort by the Dose Escalation Committee. Dose escalation will begin at dose level 1 = 420 mg.

The dose escalation will be performed for two types of associations in five separate groups :

* Group A : ibrutinib D1-D21+ R-DHAP
* Group B : ibrutinib D1-D21 R-DHAOx
* Group Abis : ibrutinib D5-D18+ R-DHAP
* Group Bbis : ibrutinib D5-D18 R-DHAOx

This dose escalation will be followed by an exploratory expansion phase in the group Bbis plus a new group including only mantle cell lymphoma (MCL) in first line patients: group C. Patients included in the Group C will receive ibrutinib in combination with R-DHAP or R-DHAOx according to the choice of the local investigator at time of inclusion of each patient.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the recommended dose of ibrutinib when administered in combination with R-DHAP (rituximab + dexamethasone + cytarabine + cisplatin) or with R-DHAOx (rituximab + dexamethasone + cytarabine + oxaliplatin) in patients with relapsed or refractory B-cell malignancies eligible for autologous stem cell transplantation (ASCT) by assessing the maximum tolerated dose (MTD) observed during the dose escalation part of the study. Assessment of the MTD will be performed by the analysis of the dose-limiting toxicities (DLTs).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with any type of relapsed or refractory B-cell lymphoma will be eligible in groups A, A bis, B and B bis (during the dose escalation and the expansion parts of the study) and untreated patients with mantle cell lymphoma will be eligible for group C (only during the expansion part of the study)
2. Each patient (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study
3. Patients eligible for autologous stem cell transplantation (ASCT) for whom R-DHAP or R-DHAOx is an acceptable therapy regarding the investigator's opinion
4. Measurable disease defined by at least one single node or tumor lesion > 1.5 cm
5. Patients who received prior therapy with at least one but no more than two lines therapies for B-Cell Lymphoma (except for patients included in group C during the expansion part of the study)
6. Aged between 18 years and 70 years (included)
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
8. Any of the following hematology values within 14 days prior to inclusion and prior to the first dose of study drug :

   1. Absolute neutrophil count (ANC) > 1,000 cells/mm3 (1.0 x 109/L) unless if bone marrow infiltration from lymphoma
   2. Spontaneous Platelets count > 75,000 cells/mm3 (75 x 109/L) within 7 days of any platelet transfusion (allowed up to 50 x 109/L if due to bone marrow infiltration from lymphoma)
9. Patients assessed as being able to receive full doses of R-DHA(P/Ox) for 3 cycles or 4 cycles for patients included in group C of the expansion phase
10. Life expectancy of ≥ 90 days (3 months)
11. Women of childbearing potential* and men who are sexually active must be practicing a highly effective method of birth control during the study and during 12 months after the end of treatments. Men must agree to not donate sperm during the study and during 12 months after the end of treatments
12. Women of childbearing potential must have a negative serum beta human chorionic gonadotropin (β-hCG) or urine pregnancy test at Screening

Exclusion Criteria:

1. Previous treatment with a BTK inhibitor
2. Patients who progressed or became refractory while on treatment with a phosphoinositide 3-kinase (PI3K) inhibitors
3. Inability to tolerate 4 courses of high dose ara-C / platin compound, especially if due to underlying comorbidities
4. History of stroke or intracranial hemorrhage within 6 months prior to the first dose of study drug
5. Major surgery, within 4 weeks prior to the first dose of study drug
6. Known bleeding diathesis
7. Condition that requires therapeutic anticoagulation with Vitamin K antagonists
8. Condition that requires treatment with a strong cytochrome P450 3A4/5 (CYP3A4/5) inhibitor
9. Any life-threatening illness, serious medical condition, laboratory abnormality, organ system dysfunction or psychiatric illness which, in the investigator's opinion, could compromise the patient's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk and that would prevent the patient from signing the informed consent form
10. Known central nervous system or meningeal involvement by lymphoma
11. Contraindication to any drug contained in these regimen
12. Known history of human immunodeficiency virus (HIV)
13. Known active Hepatitis C Virus (HCV; RNA polymerase chain reaction (PCR)-positive) or active Hepatitis B Virus infection (HBs Ag positive or DNA PCR-positive) or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics. Patients with PCR-negative for hepatitis B virus (HBV) are permitted in the study.
14. Left ventricular ejection fraction (LVEF) < 45% as determined by echocardiography or multiple uptake gated acquisition (MUGA) scan
15. Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months prior to the first dose of study drug, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
16. Any of the following biochemical values within 14 days prior to inclusion and prior to the first dose of study drug :

    1. Serum glutamic-oxaloacetic transaminase/aspartate aminotransferase (SGOT/ASAT) or serum glutamic-pyruvic transaminase/alanine aminotransferase (SGPT/ALAT) > 3.0 x upper limit of normal (ULN)
    2. Serum total bilirubin > 2.0 mg/dL (34 µmol/L), except in patients with hemolytic anemia or with Gilbert syndrome,
    3. Calculated creatinine clearance of < 50 mL /min (for patients who will have DHAOx chemotherapy) or < 70 mL/min (for patients who will have DHAP chemotherapy)
17. Patients with pre-existing ≥ Grade 2 neuropathy
18. Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the patient has been free of the disease for ≥ 3 years
19. Use of any standard or experimental anti-cancer drug therapy within 28 days prior to the first dose of study drug
20. Women who are pregnant or breastfeeding
21. Medical history of hepatic chronic disease whatever the anteriority
22. Sinusoidal obstruction syndrome (Veno-Occlusive Disease (VOD)) whatever the anteriority

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-05-26 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the incidence rate of DLTs at each dose level on cycle 1 | 21 days
  Determine the recommended phase II dose (RP2D) of ibrutinib when administered in combination with R-DHAP (rituximab + dexamethasone + cytarabine + cisplatin) or with R-DHAOx (rituximab + dexamethasone + cytarabine + oxaliplatin) in patients with relapsed or refractory B-cell malignancies eligible for autologous stem cell transplantation (ASCT) by assessing the maximum tolerated dose (MTD) observed during the dose escalation part of the study. Assessment of the MTD will be performed by the analysis of the dose-limiting toxicities (DLTs).

SECONDARY OUTCOMES:
Secondary safety endpoints | 84 days
  Study drug administration including treatment duration, average dose, dose reduction; Treatment discontinuation, study discontinuation; Adverse events, vital sign measurements, clinical laboratory measurements, and concomitant therapies.
Response Rate | 30 days after the last dose of study drug is administered
  Disease response evaluation at 3 cycles (or 4 cycles for patients with mantle cell lymphoma in first line in the expansion phase) will be used to determine the Response Rate. Response after 3 cycles (or 4 cycles) will be assessed at the end of completion of the cycles if patient received all cycles or at withdrawal
Duration of response (DoR) | from first evidence of response to the date of first documented disease progression, relapse or death from any cause, assessed up to 52 months
  Duration of response is defined as the time from first evidence of response (PR or better) to first documented disease progression, relapse or death from any cause. Patients alive and free of progression at data cut-off will be censored at the last adequate tumor assessment indicating no disease progression
Progression-Free Survival (PFS) | from the date of inclusion to the date of first observation of documented disease progression or death due to any cause, assessed up to 52 months
  PFS is defined as the time from inclusion into the study to the first observation of documented disease progression or death due to any cause. If a patient has not progressed or died, PFS will be censored at the time of last visit with adequate assessment. Patients without documented event at the time of analysis will be censored at their last follow-up date.
Time to Next Anti-Lymphoma Treatment (TTNLT) | from the date of inclusion to the date of first documented administration of any new anti-lymphoma treatment, assessed up to 52 months
  TTNLT is defined as the time from the date of inclusion to the date of first documented administration of any new anti-lymphoma treatment (chemotherapy, radiotherapy, radio-immunotherapy, immunotherapy). Patients continuing in response or who are lost to follow-up will be censored on their last visit date. Patients who died (due to any cause) before having received a new anti-lymphoma treatment will be included in the statistical analysis with death being counted as an event.
Overall Survival (OS) | from the date of inclusion to the date of death from any cause, assessed up to 52 months
  Overall survival is defined as the time from the date of inclusion to the date of death from any cause. Patients who did not die will be censored at their last follow-up date.
Pharmacokinetics profile of ibrutinib in Groups A bis and B bis | During dose escalation part, on first day of ibrutinib administration (Day 5) and on Day 15 of cycle 1 and cycle 2
  The objective is to assess the pharmacokinetic profile of ibrutinib in the presence of R-DHA(P/Ox) for groups A bis and B bis during the dose escalation part.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles SALLES, PhD, Study Chair — CHU Lyon - Sud - LYSA; Christophe BONNET, MD, Study Chair — CHU Liège - LYSA
Locations (15):
- Belgium (3):
  - Universite Catholique de Louvain Saint Luc, Brussels
  - CHU de Liège, Liège
  - CHU UCL Namur asbl, Yvoir
- France (12):
  - Centre François Baclesse, Caen
  - Hôpital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - Centre Léon Bérard, Lyon
  - CHU Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Hôpital Saint Louis, Paris
  - Centre François Magendie - Hôpital du Haut Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen